CLINICAL TRIAL: NCT06275893
Title: Phase 1b Study of IC14 in Arrhythmogenic Cardiomyopathy
Brief Title: IC14 (Atibuclimab) in Arrhythmogenic Cardiomyopathy
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study paused but may start again in the future.
Sponsor: Implicit Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACM01
Record Dates: First submitted 2024-02-06; First posted 2024-02-23 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Arrhythmogenic Right Ventricular Dysplasia; Arrhythmogenic Left Ventricular Cardiomyopathy; Arrhythmogenic Right Ventricular Cardiomyopathy 1; Arrhythmogenic Cardiomyopathy; ACM; ARVC; PKP2
Keywords: arrhythmia; cardiac genetic disorder; desmoglein mutation
MeSH Terms: conditions — Arrhythmogenic Right Ventricular Dysplasia; Arrhythmogenic Right Ventricular Dysplasia, Familial, 1; Arrhythmias, Cardiac | interventions — atibuclimab

STUDY DESIGN:
Intervention Model Description: Open-label treatment with IC14. Participant outcomes will be compared to baseline. Pharmacokinetics will be measured.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- IC14 (atibuclimab) (Experimental): IC14 (atibuclimab) 20 mg/kg intravenously every 3 weeks for 12 weeks (4 doses)
  Interventions: Biological: IC14

INTERVENTIONS:
Biological: IC14 — recombinant monoclonal antibody directed against cluster of differentiation 14 (CD14) antigen
  Other Names: (atibuclimab)

SUMMARY:
The goal of this clinical trial is to test IC14 (atibuclimab) in patients with arrhythmogenic cardiomyopathy (ACM) and who have an implantable cardoverter/defibrillator in place. ACM is also called arrhythmogenic right ventricular dysplasia (ARV) or arrhythmogenic right ventricular cardiomyopathy (ARVC). The main questions the study aims to answer are the effect of treatment on blood markers of inflammation, safety, and pharmacokinetics. There will also be measurements of myocardial imaging of C-C chemokine receptor type 2 (CCR2+) immune cells (optional), monitoring of cardiac arrhythmias using the patient's pre-existing intracardiac cardioverter/defibrillator (ICD) and a Holter monitor, electrocardiogram (ECG), echocardiogram (ECHO), and blood tests. Results will be compared to baseline; there is no inactive placebo treatment group.

Participants will be asked to undergo screening and baseline testing, then receive 4 intravenous infusions with blood measurements before and after the infusion (including 24, 48, and 72 hours and 7, 14, and 28 days). Participants will be offered specialized scanning of the heart muscle, and will be asked to provide recordings from their ICD, undergo Holter monitoring twice, and have electrocardiograms (ECG), echocardiograms (ECHO) and blood tests.

DETAILED DESCRIPTION:
This proof-of-concept study will evaluate the safety, pharmacokinetics, and preliminary efficacy of IC14 administered via IV infusion in patients with ACM.

In preclinical studies, anti-CD14 treatment prevented the development of ventricular dysfunction and cardiac damage in a mouse model of arrhythmogenic cardiomyopathy.

The objective of this study is to determine whether IC14 treatment reduces markers of inflammation and disease biomarkers in ACM patients treated with IC14. Secondary objectives are to further characterize the effect of IC14 treatment on CCR2+ cell myocardial infiltration measured by myocardial positron emission tomography (PET)/CT imaging, ventricular premature contractions (VPCs), other arrhythmias, ICD discharges, NYHA functional classification, and quality of life.

To characterize safety of IC14, the following assessments are to be performed: clinical biochemistry (safety analyses), ECG, ECHO, adverse events (AEs), serious adverse events (SAEs), and formation of anti-drug antibodies.

Finally, pharmacokinetic/pharmacodynamic parameters will be conducted. These include blood test measurements levels of the drug and its binding to its target in the serum and on cells.

This study will assign 5 patients to intravenous (IV) administration of IC14 (atibulcimab) at 20 mg/kg. The study drug will be administered every three weeks via IV infusion, for a total of 4 infusions (12 weeks of treatment).

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for the study if all of the following criteria are met:

1. Age ≥ 18 years
2. Diagnosis of arrhythmogenic cardiomyopathy and: 1) meeting the 2020 Modified Task Force Criteria as affected;
3. Left ventricular ejection fraction of ≥30%
4. Functioning implantable cardioverter/defibrillator with remote interrogation capability
5. One of the following: 1) a history of ventricular tachycardia or ventricular fibrillation (VF); 2) ≥500 ventricular premature contractions (VPCs) in 24 hours on the most recent 24-hour Holter monitor recording; or 3) C-reactive protein >=1.5 mg/mL
6. Agreement by subject, physician, and cardiologist to not change concomitant ACM medications or to conduct catheter ablation during study participation unless needed for management of life-threatening conditions
7. Capable and willing to provide informed consent
8. Capable of completing study visits
9. Females participating in the study must meet one of the following criteria:

   1. Surgically sterilized (e.g., hysterectomy, bilateral oophorectomy, or tubal ligation) for at least 6 months or postmenopausal (postmenopausal females must have no menstrual bleeding for at least 1 year) or
   2. If not postmenopausal, agree to use a double method of contraception, one of which is a barrier method (e.g., intrauterine device plus condom, spermicidal gel plus condom) until 30 days after the IC14 treatment and have negative human chorionic gonadotropin (β-hCG) test for pregnancy at Screening
10. Males who have not had a vasectomy must use appropriate contraception methods (barrier or abstinence) until 30 days after IC14 treatment

Exclusion Criteria:

A patient fulfilling any of the following criteria is to be excluded from enrollment in the study:

1. Prior myocardial infarction
2. Receiving continuous infusion of antiarrhythmic medication at time of enrollment
3. Previous major vascular intervention within 4 weeks
4. NYHA heart failure class IV, except palpitations
5. Major surgery within 6 weeks
6. Patient has participated in any study using an investigational drug or device within 30 days
7. Life expectancy of less than 1 year due to non-cardiac pathology
8. History of allergic reaction to atibuclimab (IC14) or any monoclonal antibody drug product or other CD14-derived drug product or any component used in the study (including contrast media)
9. Known severe renal (creatinine clearance <30 mL/min/m2) or hepatic insufficiency as well as alanine transaminase (ALT)/aspartate transaminase (AST) elevations ≥ 3x upper limit normal (ULN); isolated AST elevation is not considered an exclusion criterion from study participation
10. Current or planned use of continuous high-dose corticosteroids (short courses of corticosteroids are allowable)
11. Chronic immunosuppression with disease-modifying anti-rheumatic drugs (DMARDS)
12. Any clinically significant abnormality identified at the time of Screening that in the judgment of the Investigator or any sub-Investigator would preclude safe completion of the study
13. Patients who will be inaccessible due to geographic or social factors during treatment or follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety: Treatment-emergent adverse events and serious adverse events | Baseline through 14 weeks
  Treatment-emergent adverse events and serious adverse events
Safety: Incidence of anti-drug antibodies | Baseline, 4 weeks, and 14 weeks
  Incidence of anti-drug antibodies

SECONDARY OUTCOMES:
Inflammatory biomarker C-reactive protein | Baseline, 12 weeks
  Change in concentration from baseline at 12 weeks
CCR2+ Myocardial Imaging (optional) | Baseline compared to 12 weeks
  Mean change in CCR2+ cell myocardial infiltration measured by CCR2+ PET/CT imaging (standardized uptake value)
Ventricular tachycardia | Baseline compared to 12 weeks
  Number of ventricular tachycardia runs in a 7-day Holter monitor
Ventricular premature contractions | Baseline compared to 12 weeks
  Frequency of ventricular premature contractions in a 7-day Holter monitor
Sustained and non-sustained ventricular tachycardia | Baseline through 12 weeks
  Number of episodes of sustained and non-sustained ventricular tachycardia documented by ICD
Treated ventricular tachycardia | Baseline through 12 weeks
  Number of episodes of treated ventricular tachycardia (pacemaker and/or defibrillation) by ICD
Atrial premature contractions | Baseline compared to 12 weeks
  Number of atrial premature contractions in a 7-day Holter monitor
New York Heart Association (NYHA) Functional Class | Baseline compared to 12 weeks
  Change in NYHA Functional Class Questionnaire
Implantable cardioverter/defibrillator (ICD) discharges | Baseline through 12 weeks
  Frequency of ICD discharges (appropriate and/or inappropriate)
Quality-of-Life Score determined by the Kansas City Cardiomyopathy Questionnaire | Baseline compared to 12 weeks
  Change in Quality-of-Life Score determined by the Kansas City Cardiomyopathy Questionnaire, range 0 (very poor) to 65 (excellent)
Disease biomarker Troponin I | Baseline, 12 weeks
  Change in concentration from baseline at 12 weeks
Disease biomarker N-terminal B-type natriuretic peptide (NT-pro-BNP) | Baseline, 12 weeks
  Change in concentration from baseline at 12 weeks
Inflammatory biomarker interleukin (IL)1-beta | Baseline, 12 weeks
  Change in concentration from baseline at 12 weeks
Pharmacokinetics: Serum IC14 concentration versus time curve | Baseline through 14 weeks
  Area under the serum concentration versus time curve (AUC)
Pharmacokinetics: Peak serum IC14 concentration | Baseline through 14 weeks
  Peak serum IC14 concentration
Pharmacokinetics: Half life | Baseline through 14 weeks
  Half-life of serum IC14 concentration
Pharmacodynamics: Receptor Occupancy | Baseline through 14 weeks
  Measurement of monocyte membrane CD14 receptor occupancy
Pharmacodynamics: Effective Concentration 95% | Baseline through 14 weeks
  Estimation of serum concentration of IC14 to achieve 95% monocyte membrane receptor occupancy

CONTACTS AND LOCATIONS:
Overall Officials: Jan Agosti, MD, Study Director — Implicit Bioscience
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No